CLINICAL TRIAL: NCT06400992
Title: Investigation of Sky Automatic Technologies in Pediatrics
Acronym: SKY-MARVEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Advanced Bionics AG (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230143; 2023-A02351-44 (Other: ID-RCB)
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss
Keywords: Hearing Loss; cochlear implant; hearing aid; hearing device; hearing system; Simplified French Matrix Test; Noise block; background noise; target cochlear implant; pediatric cochlear implant processor
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilaterally implanted patients (Experimental): patient with two cochlear implant in each ear
  Interventions: Device: Cochlear implant processor Sky CITM M90 (CI-5295); Device: Hearing Aid, including sound processor Phonak: Sky Link M90; Diagnostic Test: French simplified matrix test (FraSimat); Behavioral: Audiologist Fitting Questionnaire; Behavioral: Patient Satisfaction Questionnaire; Behavioral: AutoSens Feedback Discussion Form
- Bimodal patients (Experimental): patient with cochlear implant in one ear and fitted with hearing aid audio in the other ear
  Interventions: Device: Hearing Aid, including sound processor Phonak: Sky Link M90; Diagnostic Test: French simplified matrix test (FraSimat); Behavioral: Audiologist Fitting Questionnaire; Behavioral: Patient Satisfaction Questionnaire; Behavioral: AutoSens Feedback Discussion Form

INTERVENTIONS:
Device: Cochlear implant processor Sky CITM M90 (CI-5295) — The Sky CI available to included patients (no procedures added) offers the AutoSense Sky OS technology with the three following programming conditions possible. This three condition are fitting and evaluated in noise 6 months after inclusion:
  1. Omnidirectional mode : no sound treatment
  2. AS Target : Autosense is active and no modifications are made by clinician
  3. AS Clinique : Autosense is active and modified by the clinician
  Arms: Bilaterally implanted patients
Device: Hearing Aid, including sound processor Phonak: Sky Link M90 — The device is fitting and programmed for home especially for the purpose research at inclusion. The Clinical map parameters will be verified according to clinical routine.
  The Sky Link offers the AutoSense Sky OS technology with the three following programming conditions possible. This three condition are fitting and evaluated in noise 6 months after inclusion:
  1. Omnidirectional mode : no sound treatment
  2. AS Target : Autosense is active and no modifications are made by clinician
  3. AS Clinique : Autosense is active and modified by the clinician
Diagnostic Test: French simplified matrix test (FraSimat) — The FraSimat speech in noise test will be tested, 6 months before inclusion in the three different fitting configurations: omni, AS clinic, AS Target. The speech will be presented from the front, noise from 180°. Noise will be presented at a fixed level of 65 dB SPL while the speech signal will be adapted to find the 50% speech reception threshold (SRT).
Behavioral: Audiologist Fitting Questionnaire — After the fitting of Hearing Aid at inclusion, the audiologist will complete a questionnaire describing the fitting and justifying fitting decisions and will collect the demographic information
Behavioral: Patient Satisfaction Questionnaire — The patient will be giving a Patient satisfaction Questionnaire, with questions regarding device and accessory use. The audiologist will go over the instructions for filling out the questionnaire at inclusion. Patients will be asked to complete the questionnaire and return it at the next visit, 6 months after inclusion.
Behavioral: AutoSens Feedback Discussion Form — 6 months after inclusion and fitting, the audiologist discusses the use of AS clinic with the subject and completes the AS questionnaire (questionnaire on the experience of using the processor in different listening situations).

SUMMARY:
The hypothesis of this research is that the AS Target setting provides the best estimate of the settings required to optimize listening in noise. As such, it is expected that speech in noise performance will be best in the AS Target condition, followed by the AS Clinic condition, and the Omni condition will be the least favourable for speech in noise performance.

DETAILED DESCRIPTION:
The ability to hear speech in noise is particularly important for children, as they are often in complex listening situations like classrooms or playgrounds. In children with hearing loss, the ability to understand speech in noise is further degraded not only by decreased audibility of speech sounds, but also additionally by the distortion spectral and temporal processing cues, and reduced binaural processing abilities. Cochlear implant manufacturers have introduced a number of technologies designed to improve speech recognition in background noise. Sound processing algorithms use a variety of strategies to facilitate listening in noise, and research has shown that these advances do lead to improved performance.

AutoSense Sky OS 3.0 (AutoSense Sky OS, AS) is an automatic auditory scene classification system specifically designed for children's typical listening situations, like classrooms and playgrounds. This technology is available in the new Sky CI M90 (Sky CI), which is the latest generation of sound processor (SP) from Advanced Bionics, designed for children.

This algorithm is also available in the Sky Link M90 hearing aid (Sky Link). This means that bimodal patients, using one Sky Link and one Sky CI can benefit from AutoSense Sky OS in addition to children with two Sky CI. The combination of the two hearing devices (HD) tested in this research, whether it be two Sky CI or one Sky CI and one Sky Link, will be referred to as the Sky Hearing System (Sky HS).

As usual in standard care, children with Sky HS can have their hearing system programmed in three ways (at the discretion of the clinician):

1. Omnidirectional mode, in which the AutoSense Sky OS is deactivated and no modifications are made by the clinician (no sound treatment)
2. AS Target, in which the AutoSense Sky OS is active and programmed with the parameters suggested by the programming software (Target) and no modifications are made by the clinician
3. AS clinic, in which the AutoSense Sky OS is active, and settings have been modified by the clinician (mixed setting).

The goal of this research is to compare speech in noise perception in each of those three possible programming conditions used in the standard care. The hypothesis of this research is that the AS Target setting provides the best estimate of the settings required to optimize listening in noise. As such, it is expected that speech in noise performance will be best in the AS Target condition.

ELIGIBILITY:
Inclusion Criteria:

* Be between 6 and 16 years of age at the time of inclusion
* Use spoken French as their primary mode of communication
* Ability to perform the Simplified French Matrix test in Noise
* Bimodal group: use the Sky CI processor or be eligible for a Sky CI processor upgrade on one side and use a contralateral hearing aid
* Bilaterally implanted group: use two Sky CI processors or be eligible for an upgrade to two Sky CI processors
* Obtain signed consent from legal guardian(s)
* Be enrolled in a health insurance plan or eligible for coverage

Exclusion Criteria:

* Severe neurological pathology identified prior to inclusion identified by MRI + /- neuro-pediatric workup
* Severe cognitive, psychiatric, or developmental disabilities identified prior to inclusion
* Family does not understand French

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Speech in noise perception (FraSimat) | 6 months
  Difference in the FraSimat score obtained with the Sky HS programmed in Omni versus the score obtained in AS Target. The scores vary from -15,0 to +15,0, the higher the score is, better is the patient's hearing comprehension.

SECONDARY OUTCOMES:
Speech in noise perception (FraSimat) | 6 months
  Difference in the FraSimat score obtained with the Sky HS programmed in AS Clinic versus the score obtained in Omni. The scores vary from -15,0 to +15,0, the higher the score is, better is the patient's hearing comprehension.
Speech in noise perception (FraSimat) | 6 months
  Difference in the FraSimat score obtained with the Sky HS programmed in AS Clinic versus the score obtained in AS Target. The scores vary from -15,0 to +15,0, the higher the score is, better is the patient's hearing comprehension.
Patient satisfaction - device | 6 months
  A patient questionnaire will be used to determine patient satisfaction with the devices. The scores vary from 0 to 10, the higher the score is better is the patient's satisfaction.
Patient satisfaction -listening | 6 months
  With the help of the audiologist, patients will discuss and rate listening quality in different listening situations. The scores vary from 1 to 5, the higher the score is better is the patient's listening quality.
Audiologist programming modifications | 6 months
  An audiologist questionnaire will be used to determine the programming modifications and decisions made by the audiologist for each individual patient. The questionnaire doesn't involve any scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LOUNDON, MD,PhD, Study Director — APHP
Locations (1):
- Audiophonology Unit of the Ear, Nose and Throat (ENT) Department ("Oto-rhino-laryngologie (ORL) et chirurgie cervico-faciale") at the Necker-Enfants Malades hospital (AP-HP)., Paris, France

IPD SHARING:
Plan to Share IPD: No